CLINICAL TRIAL: NCT06771453
Title: The GEM Trial - Genetics Education and Equity in Maternal Fetal Medicine: A Pilot Feasibility Randomized Controlled Trial to Assess Impact of a Video Education Tool (VET) on Decisional Conflict Among Prenatal Patients
Brief Title: GEM: Impact of a Video Education Tool on Decisional Conflict Among Prenatal Patients
Acronym: GEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1721550
Record Dates: First submitted 2024-11-27; First posted 2025-01-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Aneuploidy; Genetic Counseling; Informed Consent; Decisional Conflict
MeSH Terms: conditions — Aneuploidy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Prenatal Care (No Intervention): The patient will receive routine prenatal care with no video education.
- Video Educational Tool Arm (Experimental): The patient receives routine prenatal care plus video education on prenatal genetics.
  Interventions: Other: Video Educational Tool Regarding Prenatal Genetics

INTERVENTIONS:
Other: Video Educational Tool Regarding Prenatal Genetics — Video education about prenatal genetics will include content regarding aneuploidy screening and diagnostic testing options, how to make a values-based choice, and specifics of risks/benefits/limitations of each type of testing option.
  Arms: Video Educational Tool Arm

SUMMARY:
The goal of this randomized clinical trial is to assess the impact of a video educational tool on patient decisional conflict at the time when making a decision about prenatal genetic testing. The control group will receive standard prenatal care.

The secondary aims include assessing the impact of the video educational tool versus standard care on pregnant participants': perception of likelihood of having a baby affected by a genetic problem, intended plan for genetic testing, patient-provider communication, retention of prenatal genetics knowledge, and perception of genetic data privacy.

Participants will be asked to:

1. Watch video education (if randomized to this group) and complete a baseline survey at their dating ultrasound regarding knowledge of prenatal genetics, prior experiences, and demographics
2. Complete a follow up survey after seeing their prenatal care provider regarding: decisional conflict scale with respect to prenatal genetic testing decision (primary outcome), perception of likelihood of having a baby affected by a genetic problem (secondary outcome) and the type of genetic testing chosen (secondary outcome).
3. Complete a second follow up survey six to ten weeks from the second survey to assess: Provider patient communication, retention of genetics knowledge, patient recollection of testing performed, and self-reported out of pocket cost related to genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age
* Preferred language English or Spanish
* Singleton pregnancy
* No documentation of genetic screening results or counseling during this pregnancy
* Gestational age <24 weeks

Exclusion Criteria:

* Diagnosed with a fetal anomaly
* Diagnosed with known abnormal nuchal translucency test
* Diagnosed with fetal loss
* Use of a donor oocyte (egg) this pregnancy
* Prior involvement in other research study regarding prenatal genetic testing in the past two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Score on Decisional Conflict Scale (low health literacy version of the tool) | After enrollment and up to 14 days after their first obstetric appointment in that pregnancy
  The investigators will assess the decisional conflict scale score around the time when patients make a decision about prenatal genetic screening options. The resulting score ranges from 0 to 100, with 0 indicating no decisional conflict (best outcome) and 100 indicating extremely high decisional conflict (worst outcome).

SECONDARY OUTCOMES:
Perception of likelihood of having a baby affected by a genetic problem | After enrollment and up to 14 days after their first obstetric appointment in that pregnancy
  The investigators will use a Likert scale to assess patient's perception of likelihood of having a baby affected by a genetic problem (score ranges from 1 [not likely at all] to 4 [very likely]).
Percent of patients opting to pursue genetic testing | After enrollment and up to 14 days after their first obstetric appointment in that pregnancy
  The investigators will assess the percent of participants who decide to pursue screening or diagnostic genetic testing options
Patient-provider communication | Six to ten weeks from follow up survey #1
  The investigators will use a modified doctor-patient communication questionnaire to assess how patients perceived communication and comprehension of counseling with their prenatal care provider (score 0 to 8, with higher score reflecting better communication).
Retention of Prenatal Genetics Knowledge | Six to ten weeks from follow up survey #1
  The investigators will assess prenatal genetics knowledge remote from the intervention to assess retention of its content (score 0 to 12 with a higher score reflecting more knowledge). The questionnaire was created by the investigators. It is six questions that query the participants on key content highlighted in the educational intervention; the content covered is also considered standard of care to receive in counseling in routine prenatal care (for those who were not randomized to the intervention).
Perception of genetic data privacy | Six to ten weeks from follow up survey #1
  The investigators will assess on a Likert scale how important privacy of participants' own genetic data and that of their baby were in making a decision about prenatal genetic testing (score 0 to 8 with higher score reflecting more importance)

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Infants, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT06771453/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT06771453/ICF_001.pdf